CLINICAL TRIAL: NCT02131805
Title: A Multicenter Pilot Study of Electronic Skin Surface Brachytherapy for Cutaneous Basal Cell and Squamous Cell Carcinoma
Brief Title: Electronic Skin Surface Brachytherapy for Cutaneous Basal Cell and Squamous Cell Carcinoma
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Memorial Sloan Kettering Cancer Center (Other)
Collaborators: Lynn Cancer Institute (Unknown)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 14-001
Record Dates: First submitted 2014-05-05; First posted 2014-05-06 (Estimated); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Cutaneous Basal Cell; Squamous Cell Carcinoma
Keywords: skin; Brachytherapy; 14-001
MeSH Terms: conditions — Carcinoma, Squamous Cell

ARMS (1):
- Electronic Skin Surface Brachytherapy (Experimental): The patient will undergo quality of life assessment and skin imaging (ultrasonography and reflectance confocal microscopy). Brachytherapy will be performed over six outpatient visits over 2-3 weeks, on non-consecutive days. Patients will then be followed for 5 years. Reflectance confocal microscopy is optional for the participating sites.
  Interventions: Radiation: Electronic Skin Surface Brachytherapy; Behavioral: Quality of life assessment

INTERVENTIONS:
Radiation: Electronic Skin Surface Brachytherapy
Behavioral: Quality of life assessment

SUMMARY:
The purpose of this study is to assess the effectiveness of electronic skin surface brachytherapy (ESSB) for early stage basal or squamous cell carcinoma of the skin using a new device. This new device is Nucletron's Esteya Electronic Skin Surface Brachytherapy System. The investigators want to understand what effects, good and/or bad this device for delivering brachytherapy has on your skin cancer. The investigators also want to assess the safety, cosmetic results, the effects that ESSB has on quality of life and to correlate skin imaging with clinical response to ESSB.

ELIGIBILITY:
Inclusion Criteria:

* Men or women ≥ 60 years old with estimated life expectancy of ≥ 5 years
* Histopathologic diagnosis of basal or squamous cell carcinoma
* Clinical stage T1N0M0 (by AJCC 2010 criteria)

  °Basal cell carcinoma with morpheaform, sclerosing, mixed, infiltrative or micronodular features must be ≤1 cm
* Low risk pathologic features (by AJCC 2010 criteria)
* Eastern Cooperative Oncology Group (ECOG) performance status of 0-3 (Appendix C)
* Able and willing to complete the Skindex16 and Skin Cancer Index (must be able to speak English)
* Ability to provide informed consent

Exclusion Criteria:

* BCC/SCC that was previously treated (ie, recurrent BCC/SCC)
* BCC/SCC in region adjacent to or overlapping with region of prior radiotherapy
* BCC/SCC on irregular surface (ie, target area not flat)
* BCC/SCC adjacent to or overlapping with burn or scar
* BCC/SCC in area prone to trauma (including, but not limited to the skin overlying the tibia, dorsum of hands and elbow)
* BCC/SCC in area with compromised lymphatic drainage or vascular supply
* BCC/SCC within 3 cm of another treated or untreated BCC/SCC
* Inflammatory process in target area
* Collagen vascular disease (lupus, scleroderma, rheumatoid arthritis)
* Diabetes that is poorly controlled
* Genetic disorder predisposing patient to skin cancers or radiation sensitivity (basal cell nevus syndrome, xeroderma pigmentosum, ataxia telangiectasia mutans)
* Receipt of treatment with another investigational device or drug
* Receipt of drug that will affect biologic response to radiation (radiosensitizer or radioprotector)
* High likelihood of protocol non-compliance (in opinion of investigator)

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Actual)
Dates: Start 2014-05 (Actual); Primary Completion 2025-12-23 (Actual); Study Completion 2025-12-23 (Actual)

PRIMARY OUTCOMES:
efficacy of Electronic Skin Surface Brachytherapy (ESSB) | 3 years
  Efficacy will be measured by local control of the irradiated BCC/SCC three years after brachytherapy.
assess the cosmetic outcome of ESSB | 3 years
  Cosmetic outcome will be patient-reported and clinician-assessed after brachytherapy.

SECONDARY OUTCOMES:
severity of adverse events | 3 years
  (grade 1-4 adverse events). The study will use the Common Terminology Criteria for Adverse Events (CTCAE) version 4.0 for assessing toxicity related to brachytherapy.
reported quality of life | 3 years
  Patient reported health-related quality of life outcomes will be assessed using the Skindex-16 (Appendix A) and the Skin Cancer Index (Appendix B).

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Barker, MD, Principal Investigator — Memorial Sloan Kettering Cancer Center
Locations (8):
- United States (8):
  - Boca Raton Regional Hospital, Boca Raton, Florida
  - Memorial Sloan Kettering Basking Ridge (Consent only), Basking Ridge, New Jersey
  - Memorial Sloan Kettering Monmouth (Consent only), Middletown, New Jersey
  - Memorial Sloan Kettering Bergen (Consent only), Montvale, New Jersey
  - Memorial Sloan Kettering Commack (Consent only), Commack, New York
  - Memorial Sloan Kettering Westchester (All Protocol Activities), Harrison, New York
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Memorial Sloan Kettering Nassau (Consent only), Uniondale, New York

REFERENCES:
- See also: Memorial Sloan Kettering Cancer Center — http://www.mskcc.org/